CLINICAL TRIAL: NCT06488833
Title: Evaluation of First Year Implementation of Komtü Programme to Improve Children's Emotional Well-being in Pre-school and Primary School.
Brief Title: Evaluation of First Year Implementation of Komtü Programme to Improve Emotional Well-being in School.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Autonoma de Barcelona (Other)
Collaborators: Nous Cims Private Foundation (Unknown)
Responsible Party: Principal Investigator, Sergi Ballespí, Ph.D., Principal Investigator, Universitat Autonoma de Barcelona
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023 DI 00057
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Psychological Well-Being; Mental Health Wellness
Keywords: Psychological Well-being; Emotional Well-being; Emotional Health; School Intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-post design with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Komtü Programme (Komtü) (Experimental): The Komtü is a programme that aims to enhance the well-being and the emotional support of children by providing training and support to the entire school community, with a particular focus on teachers.
  The Komtü programme comprises two distinct phases: the first, the Implementation Phase, is conducted over a period of three school years. During this phase, a specialist visits the school twice a week during the 1st and 2nd school years, and once a week during the 3rd school year. Some actions take place during this phase. For example, the specialist will provide training with reflective practice exercises, healing spaces and support for teachers and will also provide coaching for the school management team.
  The second phase, the Sustainability Phase, is also conducted over three school years. This phase is designed as a follow-up phase, which is meant to ensure the continuity of the programme at the school even in the absence of the specialist's weekly visits from the centre.
  Interventions: Behavioral: Komtü Programme (Komtü)
- Komtü Training and Reflective Practice (Experimental): This is a different version of the Komtü Programme that aims to enhance the well-being and the emotional support of children.
  In Komtü Training and Reflective Practice, the Implementation Phase is modified. The 1st school year, the specialist will only provide training with reflective practice exercises. This means, the other actions that are usually carried out by the programme will not be offered.
  In contrast to the original version, this would reduce the cost of the intervention and allow a greater number of schools to participate in the programme, as the specialist would have the time to intervene in more centres. It has been decided to prioritise training with reflective practice exercises as it is the core component that gives meaning to the functioning of the other activities that are developed throughout the programme.
  Interventions: Behavioral: Komtü Training and Reflective Practice
- Control group or Treatment as usual (TAU) (No Intervention): The school year will be developed as normal.

INTERVENTIONS:
Behavioral: Komtü Programme (Komtü) — Mainly, 4 actions will take place:
  * Training with reflective practice exercises. This is a 32-hours group training involving 21 sessions that last 60 minutes and 11 hours of inter-sessions work. The contents of the training will be 5 of the 10 total blocks of Komtü training: Block 1: Meeting, observing and listening; Block 2: Neuroscience applied in the educational context; Block 3: High- quality relationships; Block 4: Conflict management; Block 5: Boundary management
  * Healing spaces to generate a collective restorative experience, offering tools that facilitate emotional management
  * Individual support for teachers to offer them resources, tools, and intervention strategies to help improve educational practice and the emotional and relational well-being of the school community
  * Coaching for the school management team to help them establish some objectives together and offer them the necessary resources and tools so that they can achieve them successfully.
  Other Names: Komtü
  Arms: Komtü Programme (Komtü)
Behavioral: Komtü Training and Reflective Practice — This is a 32-hours group training involving 21 sessions that last 60 minutes and 11 hours of inter-sessions work. The contents of the training will be 5 of the 10 total blocks of Komtü training: Block 1: Meeting, observing and listening; Block 2: Neuroscience applied in the educational context; Block 3: High- quality relationships; Block 4: Conflict management; Block 5: Boundary management
  No other actions will take place in this group.
  Arms: Komtü Training and Reflective Practice

SUMMARY:
Objectives: (1) To analyse the benefits of Komtü Programme implementation in children's and teachers' well-being (primary outcomes); (2) to analyse the benefits of Komtü Programme implementation in teacher's assertiveness, mentalization and self-efficacy (secondary outcomes). (3) and to analyse the benefits of Komtü Programme implementation according to children's prosocial behaviour, self-esteem and mentalization (secondary outcomes).

Participants: Teachers will be placed in one of the 3 groups, according to the school's support needs they work at. In this case, randomization would not be possible in the allocation process. In one of the interventions, the participants will receive the planned actions for the first school year of the Komtü Programme. In the other intervention, the participants will only receive the training and the reflective practice planned for the Komtü. The last group will complete the school year as usual (TAU, control group).

Comparisons: Researchers will compare all 3 groups among them to see to what extent:

* Komtü Programme shows efficacy in fostering children's well-being compared with the training and TAU (control group).
* Komtü Programme shows efficacy in fostering teachers' well-being compared with the training and TAU (control group).
* Training and reflective practice shows efficacy in fostering children's well-being compared with TAU (control group).
* Training and reflective practice shows efficacy in fostering teachers' well-being compared with TAU (control group).

And as for the secondary outcomes, researchers will also compare all 3 group to observe possible inter-group differences.

DETAILED DESCRIPTION:
Context: Lately, mental health has become an important issue of global priority, especially when it comes to child and youth population. Acting during this stage of life is crucial, as the symptomatology of some mental disorders present in adulthood could start before the age of 14 in 33.3% to 50% of cases. It seems that schools could be a great context to foster mental health, as children spend most of the day hours there. At school, children not only acquire academic knowledge, they also learn emotional and social competencies and, in this process, teachers can become a model for them. However, most of the school programmes that aim to enhance children's well-being are directly implemented with children, and few programmes are designed to work with teachers. Furthermore, when implementing a school programme, it is not usual to have a specialist within the school centre, that addresses teacher's worries and accompanies them through the programme completion. That is why Nous Cims Private Foundation decided to create the Komtü programme, which aims to impact children's well-being by accompanying teachers during 3 school years by a specialist that visits the centre twice a week. As this programme is relatively new, the researchers in this study intend to: (1) analyse the benefits of Komtü programme and, considering that this is a long-term programme, (2) the investigators want to study the effectiveness of a more cost-efficient approach by only implementing the training and reflective practice associated with the programme.

Methodology: 8-month 3-armed quasi-experimental pre-post design with control group.

Measures Operationalization: It is expected that Komtü programme could benefit teachers who receive the intervention and their students, since they share a lot of classroom time. Teacher benefits are expected in terms of higher emotional well-being (primary outcome) but also in terms of higher sense of self-efficacy, higher assertiveness and improved mentalizing capacities (secondary outcomes). Children benefits are expected in terms of higher emotional well-being (primary outcome) but also in terms of mentalization, prosocial behaviour and self-esteem (secondary outcomes). We will also consider teachers' burnout and faculty trust as process outcomes since they can impact teacher's well-being.

Statistical Analyses: The analysis will encompass all participants, with the utilization of multiple imputation techniques to address any missing data. Estimation of parameters, accounting for the specific statistical assumption of each model and the data's characteristics, will be carried out using general linear modelling adjusting for baseline values. Various Stata packages will be employed to execute these models, primarily SPSS and jamovi. Concerning statistical power, a sample size of 90 teachers (30 per arm) and 180 students (90 per arm) has been proposed as the minimum required to detect a medium effect size (d=0.50) -in case of teachers- and small effect size (d =0.30) -in case of students- in the design comprising 3 arms, 2 repeated measures (pre-post), and a power level of 0.80.

ELIGIBILITY:
Inclusion Criteria:

* Teachers at public school (6 y.o. - 12 y.o.) or preschool (3 y.o. - 6 y.o.) in active
* Students from 4th, 5th and 6th grade of Primary School (9 - 12 y.o.)
* Understanding Catalan
* Written Informed Consent

Exclusion Criteria:

* Teachers at private or charter schools.
* Teachers at rural schools.
* Preschool students (3-y.o. - 6 y.o.) and students from 1st, 2nd and 3rd grade of Primary School (6 y.o. - 8 y.o.).
* Schools that already have any training/knowledge related to emotional support or emotional intelligence.

Ages: 9 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Stirling Children's Well-Being Scale (SCWB) | Through study completion, an average of 8 months
  This is a 15-item scale commonly used to measure children's happiness in the last 2 weeks. Items are scored from '1 = Never' to '5 = All the time'. The score ranges from 15 to 75. A higher score means more happiness (better outcome).
Child Well-being Level (CWBL) | Through study completion, an average of 8 months
  This is Likert's 7-point scale to assess the child's level of happiness compared with other children of the same age. It is responded by children. It ranges from '1 = Very less happy' to '7 = Very happier'. A higher score means more happiness (better outcome).
Child Well-being Level - Teacher's version (CWBL-T) | Through study completion, an average of 8 months
  This is Likert's 7-point scale to assess the child's level of happiness compared with other children of the same age. It is responded by teachers. It ranges from '1 = Very less happy' to '7 = Very happier'. A higher score means more happiness (better outcome).
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Through study completion, an average of 8 months
  This is a 14-item scale commonly used to measure mental well-being in general population in the last 2 weeks. Items are scored from '1 = None of the time' to '5 = All of the time'. The score ranges from 14 to 70. A higher score means more well-being (better outcome).
Teacher's Subjective Well-being Scale (TSWBS) | Through study completion, an average of 8 months
  This is a 8-item scale used to measure teacher's subjective well-being according to 2 sub-scales: teaching efficacy (4 items) and school connectedness (4 items). Items are scored in 4-points Likert scale ranging from '1 = Almost never' to '4 = Almost always'. The score ranges from 8 to 32. A higher score means more well-being (better outcome).

SECONDARY OUTCOMES:
Bar-On Emotional Quotient Inventory: Youth Version (BarOn EQ-i: YV) | Through study completion, an average of 8 months
  BarOn's scales of intra-personal (6 items) and inter-personal (12 items) scales, which are scored in 4-points Likert scales ranging from '1 = Never' to '4 = Always'. The indicated subscales ranges are 4-24 and 12-48, respectively. A higher score indicates higher emotional intelligence (better outcome).
Self-Other Mentalization Scale (SOMS) | Through study completion, an average of 8 months
  These are two Likert's 5-point scales to assess the child's mentalization compared with other children of the same age. It is responded by their teachers. It ranges from '1 = Far less than others' to '5 = Far more than others'. A higher score means more mentalization (better outcome).
Rosenberg's Self-Esteem Scale - Child version (RSES-C) | Through study completion, an average of 8 months
  This is a gold standard measure of self-esteem using 10 items which are scored from '1 = Totally agree' to '4 = Totally disagree'. After inverting the total score, which ranges from 10 to 40, a higher score means higher self-esteem (better outcome).
Strengths and Difficulties Questionnaire (SDQ) | Through study completion, an average of 8 months
  Prosocial SDQ scale (5 items), which are scored in 3-point Likert scales ranging from '0 = Not true' to '2 = Certainly true'. The indicated subscale range is 0 from 10. A higher score indicates more prosocial behaviour (better outcome).
Mentalization Scale (MentS) | Through study completion, an average of 8 months
  This is a 28-item scale to assess 3 dimensions of mentalization: self-related mentalization, other-related mentalization and motivation to mentalize. Items are scored from '1 = Completely incorrect' to '5 = Completely correct'. The indicated subscales scores can range from 8 to 64, from 10 to 50 and from 10 to 50, respectively. A higher score means more mentalization (better outcome).
Teacher Self-Efficacy Scale - Short Form (TSES-S) | Through study completion, an average of 8 months
  This is a 12-item scale to assess teacher's self-efficacy according to 3 subscales: efficacy in student engagement (4 items), efficacy in instructional strategies (4 items) and efficacy in classroom management (4 items). Items are scored from '1 = Nothing' to '9 = A Great Deal'. The indicated subscales range is 4-36. A higher score means more teachers' sense of efficacy (better outcome).
Self-reports of Assertive Behaviour: Attitudes and Values in Social Interactions (ADCAs) | Through study completion, an average of 8 months
  This is a 35-item scale to assess auto-assertiveness (20 items) and hetero-assertiveness (15 items) in general population. It also contains a specific form to assess teacher's assertiveness in classroom interactions. Items are scored from '1 = Never or Hardly ever' to '4 = Always or Most of the time'. The indicated subscales ranges are 20-80 and 15-60, respectively. A higher score means more assertiveness (better outcome).

OTHER OUTCOMES:
Maslach Burnout Inventory - Educators Survey (MBI-ES) | Through study completion, an average of 8 months
  This is a 22-item inventory that assesses burnout for people working in an educational setting according to 3 dimensions: emotional exhaustion (9 items), depersonalization (5 items) and personal accomplishment (8 items). Items are scored from '0 = Never' to '6 = Every day'. The indicated subscales ranges are 0-54, 0-30 and 0-48, respectively. In emotional exhaustion and depersonalization subscales, a higher score means more emotional exhaustion and depersonalization, respectively (worse outcome). In personal accomplishment, a higher score means more personal accomplishment (better outcome).
Omnibus Trust Scale | Through study completion, an average of 8 months
  This is a 26-item scale that assesses teachers' trust in principals, parents, students and colleagues. It is divided into three subscales: faculty trust in the principal (8 items), faculty trust in colleagues (8 items) and faculty trust in clients, which includes parents and students (10 items). Items are scored from '1 = Strongly disagree' to '6 = Strongly agree'. The indicated subscales ranges are 8-48, 8-48 and 10-60, respectively. A higher score means more faculty trust (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Ballespí, PhD, Study Director — Universitat Autònoma de Barcelona (UAB); Elena Gervilla, PhD, Study Director — Universitat de les Illes Balears (UIB)
Locations (1):
- Nous Cims Private Foundation, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Komtü Programme website (English not available) — http://www.komtu.org/es/
- See also: Nous Cims Private Foundation website (English version) — http://www.nouscims.com/en/